CLINICAL TRIAL: NCT03111264
Title: Building Blocks for Healthy Preschoolers: Child Care and Family Models
Brief Title: Building Blocks for Healthy Preschoolers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 Closures & Lockdown
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00065933; 1R01DK107761-01 (NIH)
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Obesity
Keywords: Overweight; Obesity; Prevention; Children; Childcare; Physical Activity; Nutrition; Wellness; Environment; Intervention; Feeding
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Motor Activity | interventions — Mov10l1 protein, mouse

STUDY DESIGN:
Intervention Model Description: The investigators will examine the impact of the teacher-led CHAMP intervention individually and combined with a CHAMP+ parenting intervention versus control on child BMI z-score, food tasting, food preferences and knowledge, gross motor skills, and physical activity.
Who Masked: Participant
Masking Description: One third of recruited childcare centers (control) will not receive any intervention (CHAMP nor CHAMP+). The remaining two-thirds of the recruited centers will receive the CHAMP intervention, of those, one third will also receive the CHAMP+ parenting intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHAMP group (Experimental): Childcare centers randomly assigned the CHAMP group will receive an intervention that promotes physical activity in the classroom by developing gross motor skills through movement and enhances the nutritional environment in the centers by exposing preschoolers to new foods.
  Interventions: Behavioral: CHAMP
- CHAMP+ group (Experimental): These childcare centers, also randomly assigned, will have the same intervention as the CHAMP group in addition to a parenting intervention that promotes wellness and healthy behaviors within families.
  Interventions: Behavioral: CHAMP; Behavioral: CHAMP+
- Control (No Intervention): This group will not receive theCHAMP intervention at the childcare center nor will this group receive the CHAMP+ parenting intervention.

INTERVENTIONS:
Behavioral: CHAMP — The CHAMP only group intervention is based on "Food Friends & Mighty Moves", a nutritional program designed to introduce new foods over the course of 12 weeks to preschoolers to create positive eating experiences. In conjunction with the nutritional program, the intervention also consists of an 18 week physical activity program designed to develop gross motor skills.
  Arms: CHAMP group; CHAMP+ group
Behavioral: CHAMP+ — The CHAMP+ component is comprised of a curriculum of parenting, wellness, physical activity, and feeding in the home environment. The CHAMP+ intervention will span over the course of the CHAMP intervention.
  Arms: CHAMP+ group

SUMMARY:
Pediatric obesity, a defining health problem of the century, leads to long-term health disparities. This application evaluates strategies to prevent health disparities early in life by developing environmental wellness-related interventions focused on child-care center staff and families.

Childcare centers provide an excellent opportunity to build healthy dietary and physical activity lifestyle habits and avoid the rapid weight gain that leads to health disparities. Building on a statewide survey among childcare centers and a pilot evaluation of an environmental intervention, this 3-cell randomized trial evaluates the impact of a staff-led wellness intervention and a staff-led and family-focused intervention, against a control condition.

DETAILED DESCRIPTION:
The intervention trial will be conducted in 48-55 childcare centers throughout Maryland, enrolling 864 children age 30-54 months from childcare centers serving low-income families. The aims are:

1. to examine the impact of the wellness intervention individually and combined with the family intervention versus control on BMI z-score, food preferences and knowledge, and physical activity among children
2. to examine the sustainability of the interventions
3. to examine whether changes in outcomes measures for children's BMI z-score, gross motor skills, food preferences and knowledge, and physical activity are mediated by changes in the childcare staff wellness-related attitudes and behaviors and/or parent wellness-related attitudes and behaviors (exploratory).

Findings from the trial will inform programs and policies in childcare centers to prevent obesity and reduce disparities, and will be disseminated locally, regionally, and nationally through conferences, information briefs, social media, and peer-reviewed journal articles. The overall objective is to promote statewide strategies that reduce pediatric obesity and the long-term health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Preschooler 30-54 months
* Caregiver and childcare staff must be at least 18 years old
* Childcare center staff members willing to participate
* Licensed childcare centers serving low-income communities
* Children attending participating childcare centers (at least 3 days per week)

Exclusion Criteria:

* Caregivers and staff who do not speak or read English
* Childcare staff and preschoolers with health problems that would interfere with participation in physical activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1943 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change of BMI Z-score for preschoolers | Baseline to 6 month (Midline) Follow-up or 1 year (Post Intervention) Follow-up
  Measured weight and height for the preschoolers, calculated as age and gender-specific BMI Z-score

SECONDARY OUTCOMES:
Change of Physical Activity for preschoolers and childcare center staff | Baseline to 6 month (Midline) Follow-up or 1 year (Post Intervention) Follow-up
  Moderate to Vigorous Physical Activity (MVPA) based on anthropometrics
Change in Gross Motor Skills | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up
  Measured by Test of Gross Motor Development-2
Change in Preschoolers to try new foods | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up
  Measured by Food Neophobia Scale (Caregiver report)
Change in Preschoolers to try new foods | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up
  Measured by Fruit & Vegetable Knowledge & Preference Test
Change in Preschoolers to try new foods | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up
  Measured by Food Tasting Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Growth and Nutrition Division, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowalski AJ, Armstrong B, Trude ACB, Arbaiza R, Czinn A, Bellows LL, Johnson SL, Wang Y, Hager ER, Black MM. Creating healthy habits for Maryland preschoolers (CHAMP): a cluster-randomized controlled trial among childcare centers. Int J Behav Nutr Phys Act. 2025 Dec 10;22(1):156. doi: 10.1186/s12966-025-01824-6. PMID 41372951
- [Derived] Rahmaty Z, Johantgen ME, Storr CL, Wang Y, Black MM. Preschoolers BMI: Associations with Patterns of Caregivers' Feeding Practices Using Structural Equation Models. Child Obes. 2023 Apr;19(3):169-178. doi: 10.1089/chi.2022.0026. Epub 2022 Jun 1. PMID 35649202
- [Derived] Armstrong B, Trude ACB, Johnson C, Castelo RJ, Zemanick A, Haber-Sage S, Arbaiza R, Black MM. CHAMP: A cluster randomized-control trial to prevent obesity in child care centers. Contemp Clin Trials. 2019 Nov;86:105849. doi: 10.1016/j.cct.2019.105849. Epub 2019 Sep 13. PMID 31525490